CLINICAL TRIAL: NCT07166926
Title: Mobile Pediatric Thoracic and Abdominopelvic Computed Tomography (CT)
Brief Title: Pediatrics Mobile CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00118586
Record Dates: First submitted 2025-09-09; First posted 2025-09-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Abdominal Imaging; Pediatric Imaging
Keywords: SOMATOM On.site

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Mobile CT for pediatric patients in NICU, CVICU, and PICU (Other): Pediatric patients in NICU, CVICU, and PICU who are too ill to transport to the radiology department; could benefit from imaging for diagnosis and care. Advanced imaging modalities like CT can provide critical insights for monitoring pediatric patients with certain conditions.
  Interventions: Device: Mobile CT

INTERVENTIONS:
Device: Mobile CT — SOMATOM On.site

SUMMARY:
A special kind of CT scanner that can move around (called a mobile CT) is already approved by the FDA to take pictures of adult and pediatric heads. This study wants to see if the same machine can safely take pictures of the chest and belly (abdomen) in children. This may benefit pediatric patients who may need a CT but are otherwise unable to be safely transported to the radiology department.

ELIGIBILITY:
Inclusion Criteria:

* Patient <5 years of age or meeting size criteria to fit into the CT gantry and field of view (35 cm gantry aperture, 26 cm field of view).
* Patients who would benefit from cross-sectional imaging (CT) of the chest and/or abdomen and pelvis, based on severity and anticipated progression of their disease, as determined by their primary treatment team or recommended by a consultant team.
* Patients who are deemed clinically unsafe to travel based on medical conditions as determined by their primary treatment team.

Exclusion Criteria:

* Size precludes safe operation of the CT gantry
* Unable to consent and parent/guardian unable to consent.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Images With Good or Acceptable Quality | From enrollment to interpretation of the scan (up to approximately 48 hours)
  Image quality will be considered good/acceptable if there is a clinical report. Otherwise it is unacceptable.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No